CLINICAL TRIAL: NCT01224912
Title: Phase 3 Study of Internet-based Self-help for Insomnia: Factors That Are Associated With Success of the Intervention
Brief Title: Internet Delivered Self-Help CBT for Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Utrecht University (Other)
Responsible Party: Utrecht University, Utrecht University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UU-vandenBout-2
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Insomnia
Keywords: Insomnia; Intervention; Self-help; Internet
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Internet Deliviered CBT for Insomnia (Experimental): Cognitive behavioral self-help method for insomnia via the Internet
  Interventions: Behavioral: Cognitive Behavioral Treatment

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment — The techniques used throughout the self-help manual are all effective in reducing insomnia: 1) Stimulus control: patients should only go to bed when sleepy, use the bed and bedroom for sleep (and sex) only, maintain a regular rising time, avoid daytime naps and get out of bed and go into another room when unable to fall asleep within 15-20 minutes (return only when sleepy). 2) progressive muscle relaxation. 3) sleep hygiene education (improving health and environmental factors that affect sleep). 3). Sleep restriction, whereby participants will stay only the time in bed that they sleep. 4) cognitive therapy to challenge and dispute incorrect and unhelpful thoughts about sleep (e.g. I must sleep at least 8 hours, otherwise I'll be a wreck tomorrow).

SUMMARY:
The object of this study is to determine variables associated with therapy-success of a cognitive behavioral self help intervention for insomnia. In this study all participants receive an online self-help CBT manual consisting of information (psycho-education) about sleep and cognitive-behavioural exercises. Adult persons with insomnia will be invited via a popular scientific website to fill out online questionnaires. Participants will be measured 4, 16, and 40 weeks after intervention with the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia
* Access to the internet

Exclusion Criteria:

* Alcohol or substance abuse
* Being suicidal
* Sleep apnea
* Schizophrenic or having a psychosis disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Sleep diary | baseline
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Day ratings.
Sleep diary | 4-week follow-up
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Day ratings.
Sleep diary | 18-week follow-up
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Day ratings.
Sleep diary | 48-week follow-up
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Day ratings.

SECONDARY OUTCOMES:
Anxiety | Baseline
  Measured with the HADS
Anxiety | 4-week follow-up
  HADS
Anxiety | 18-week follow-up
  HADS
Anxiety | 48-week follow-up
  HADS
Depression | Baseline
  CES-D
Depression | 4 week follow-up
  CES-D
Depression | 18-week follow-up
  CES-D
Depression | 48-week follow-up
  CES-D
Sleep medication | Baseline
  Sleep medication as measured by the sleep diary
Sleep medication | 4-week follow-up
  Sleep medication as measured by the sleep diary
Sleep medication | 18-week follow-up
  Sleep medication as measured by the sleep diary
Sleep medication | 48-week follow-up
  Sleep medication as measured by the sleep diary
Insomnia Severity | Baseline
  Insomnia Severity Index
Insomnia severity | four-week follow-up
  Insomnia Severity Index
Insomnia severity | 18-week follow-up
  Insomnia Severity Index
Insomnia severity | 48-week follow-up
  Insomnia Severity Index

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Lancee, MSc, Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Popular scientific website about insomnia — http://www.insomnie.nl